CLINICAL TRIAL: NCT04181944
Title: Qualitative Survey of Potential Exercise Activity in Adults With Sickle Cell Anemia (SCA)
Acronym: SCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCDFit
Record Dates: First submitted 2019-11-20; First posted 2019-12-02 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Cardiovascular Diseases; Sickle Cell Disease; Exercise
MeSH Terms: conditions — Cardiovascular Diseases; Anemia, Sickle Cell; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Treatment Group (Experimental)
  Interventions: Other: Exercise Treatment Group

INTERVENTIONS:
Other: Exercise Treatment Group — be specific

SUMMARY:
The purpose of this study is to assess the potential interventions of exercises in adults with sickle cell anemia (SCA) and cardiopulmonary disease; only including the more severe genotypes of sickle cell disease.

DETAILED DESCRIPTION:
Sickle cell disease is an inherited blood disorder that affects approximately 100,000 people in the United States. People living with sickle cell disease have numerous complications that cause significant morbidity and mortality such as painful episodes of vasoocclusion, acute chest syndrome, stroke, end organ damage, and early death. Unfortunately, their lifespan remains markedly shorter than the general population and this had not dramatically changed in the last 2 decades. Adults, are now not dying primarily from infections and sickle cell disease related complications, but cardiopulmonary disease is a leading cause of death. The etiology of cardiopulmonary disease in sickle cell disease is unclear but studies suggest that microvascular hypoxia, inflammation and endothelial dysfunction play a major role in the pathogenesis. In the general population, exercise reduces cardiovascular complications, pulmonary exacerbations, and decreases cardiovascular death. However, exercise used as primary or secondary prevention in sickle cell disease for cardiopulmonary disease has not been explored. Evidence shows that exercise in sickle cell disease can decrease oxidative stress, lower blood viscosity, and increase nitric oxide levels in both human and mouse models, but there remains some concern that high-intensity training in sickle cell disease may trigger vaso-occlusive crisis and adverse outcomes. However, multiple recent studies show that moderate intensity exercise can be safely performed in adults with sickle cell disease. Currently, providers lack evidence-based knowledge to inform the quantity and quality of regular exercise training that is safe but also improves cardiovascular outcomes in sickle cell disease. In addition, data does not exist on the feasibility and adherence of home-based training regimens in adults with sickle cell disease. Only one study has explored the feasibility and adherence in children. This study will be a qualitative assessment of potential interventions of exercises in adults with sickle cell anemia, only including the more severe genotypes of sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with a known diagnosis of sickle cell anemia
* Subject (and, parental/legal representative, when applicable) must understand and voluntarily sign a consent form and complete an interview

Exclusion Criteria:

- Subjects who does not meet the inclusion criteria above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-06-14 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Specific exercise regimen for those living with sickle cell disease | One year
  100 participants with sickle cell disease exercise preference based on the survey results, decrease the severity of cardiovascular disease in patients with sickle cell disease

CONTACTS AND LOCATIONS:
Overall Officials: Foluso J Ogunsile, MD, Principal Investigator — Memorial Healthcare System
Locations (1):
- Memorial Healthcare System, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No
To be determined